CLINICAL TRIAL: NCT00426205
Title: GM-CSF Secreting Leukemia Cell Vaccinations After Allogeneic Non-myeloablative Peripheral Blood Stem Cell Transplantation in Patients With Advanced Myelodysplastic Syndrome or Refractory Acute or Advanced Chronic Myeloid Leukemia
Brief Title: GM-CSF Vaccinations After Allogeneic Blood Stem Cell Transplantation in Patients With Advanced Myeloid Malignancies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Vincent T. Ho, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 04-023
Record Dates: First submitted 2007-01-23; First posted 2007-01-24 (Estimated); Last update posted 2022-02-11 (Actual); Status verified 2022-01

CONDITIONS: Myelodysplastic Syndrome RAEB-I or RAEB-II; Refractory Acute Myeloid Leukemia; Refractory CML Myeloid Blast Crisis
Keywords: GM-CSF; GVAX; Cancer vaccine; blood stem cell transplantation; MDS; AML; CML
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: GM-CSF secreting leukemia vaccine — Vaccine given subcutaneously or intradermally on the leg, arm, or abdomen 6 times. The first three vaccines will be given once a week for three weeks. The last three vaccines will be given once every other week for three doses.

SUMMARY:
The purpose of this study is to investigate whether the addition of a vaccine after participants reduced intensity transplant will be safe and beneficial. The vaccine used in this trial, called GVAX, will be made from the participants own leukemia cells, and will be given between 1-4 months after transplant. In recent years, researchers have discovered that GVAX vaccine made from the patient's own cancer calls that have been engineered in the laboratory to produce a protein called GM-CSF, can be effective in stimulating a powerful immune response specific to that cancer.

DETAILED DESCRIPTION:
* This trial can be divided into three phases: 1) Pre-transplant phase; 2) Reduced intensity transplant phase; 3) Vaccination phase.
* Pre-transplant phase: Once a suitable donor has been identified, the participant will undergo a battery of standard pre-transplant tests and procedure to collect their leukemia cells for vaccine generation. Blood tests, heart function test, pulmonary function test, tuberculosis test, bone marrow aspirate and biopsy, and leukemia cell collection through leukapheresis.
* Allogeneic reduced intensity stem cell transplant phase: The transplant phase of the study will begin when the participant is admitted to the hospital to receive the chemotherapy and stem cell transplant. The minimum duration of hospitalization for the procedure is approximately 8 days. In the week before the participant receives the stem cells, they will be treated with chemotherapy through a central line. The goal of chemotherapy is to both control the cancer and suppress the immune system so that the body will not reject the donor stem cells.
* Just prior to and immediately following the infusion of stem cells, participants will receive medications to help prevent graft-versus-host disease (GVHD), a common complication of transplant where the donor's immune cells attack the body. After the transplant, participants will also take antibiotic medication to help prevent possible infections.
* Sargramostim (GM-CSF, leukine), a white blood cell growth factor, will be given daily subcutaneously starting the day after the stem cell transplant until blood counts have recovered.
* After the stem cell infusion, participants will be examined and have blood tests weekly for 1 month. Between 30-45 days after the transplant, a bone marrow biopsy will be performed to assess the status of the disease and to look for evidence of the donor's cells in the bone marrow.
* Vaccination Phase: After the bone marrow biopsy 30-45 days after the transplant, the participant will begin to receive the vaccinations. The vaccine will be administered subcutaneously and intradermally on the arm, leg, or abdomen 6 times over a period of 9 weeks. The first 3 vaccinations will occur once a week for 3 consecutive weeks, and the last 3 vaccines will be given once every other week over 6 weeks. All vaccinations may be given as an outpatient in the clinic. During this period of time, participants will be closely monitored on a weekly basis to monitor for side effects. Before the first and after the fifth and sixth vaccinations, a small amount of the participants leukemia cells will be injected under the skin to see if the immune system will react against it and cause redness and swelling.
* About 4 weeks after the last vaccination (6th), a bone marrow aspirate and biopsy will be performed to assess the status of the disease.
* After the 1st and 5th vaccinations, a skin biopsy will be performed to assess for response at the vaccine site. These biopsies are relatively simple outpatient procedures.

ELIGIBILITY:
Inclusion Criteria:

* AML, MDS-RAEB or RAEB-T, CML, myeloid blast crisis not in remission or CML accelerated phase. Subjects must have > 5% blasts in bone marrow or peripheral blood prior to admission for transplant.
* HLA 6/6 matched related or unrelated donor available
* ECOG Performance Statue 0-2
* 18 years of age or older

Exclusion Criteria:

* Uncontrolled infection
* Leukemia with active CNS involvement
* Serum creatinine greater than 2.0 mg/dl
* ALT or AST greater than 3 x ULN
* Total bilirubin greater than 2.0 mg/dl
* Positive HIV or HTLV-1 serology
* Prior allogeneic stem cell transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2004-06; Primary Completion 2007-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Feasibility as measured by ability to generate sufficient vaccine, and ability for this patient population to initiate vaccination between day 30 to day 45 after transplant. | 3 years

SECONDARY OUTCOMES:
Safety of GVAX vaccination as measured by grade III-IV acute GVHD, and CTC grade 3 or higher non-hematologic toxicity | 3 years
biologic activity of GVAX vaccination | 3 years
disease free and overall survival.

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Ho, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States

REFERENCES:
- [Background] Ho VT, Vanneman M, Kim H, Sasada T, Kang YJ, Pasek M, Cutler C, Koreth J, Alyea E, Sarantopoulos S, Antin JH, Ritz J, Canning C, Kutok J, Mihm MC, Dranoff G, Soiffer R. Biologic activity of irradiated, autologous, GM-CSF-secreting leukemia cell vaccines early after allogeneic stem cell transplantation. Proc Natl Acad Sci U S A. 2009 Sep 15;106(37):15825-30. doi: 10.1073/pnas.0908358106. Epub 2009 Aug 26. PMID 19717467